CLINICAL TRIAL: NCT00881686
Title: Study of Myocardial Protection in Pediatric Cardiac Surgery With Adenosine Preconditioning
Brief Title: Myocardial Protection With Adenosine Preconditioning
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Zhenxiao Jin, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: xinzangwaike0002
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2009-04-15 (Estimated); Status verified 2009-03

CONDITIONS: Heart Defects, Congenital; Cardiac Surgical Procedures; Myocardial Reperfusion Injury; Adenosine
Keywords: Ischemic Preconditioning, Myocardial; Adenosine
MeSH Terms: conditions — Heart Defects, Congenital; Myocardial Reperfusion Injury | interventions — Adenosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- adenosine (Experimental): Adenosine will be administered intravenously before surgery
  Interventions: Drug: adenosine

INTERVENTIONS:
Drug: adenosine — 1.5mg/Kg adenosine will be administered intravenously before surgery

SUMMARY:
Adenosine has been proved to be an important mediator of myocardial protection induced by ischemic preconditioning. The hypothesis of this study is that adenosine preconditioning can provide additional myocardial protection in the setting of pediatric open heart surgery with cardioplegia and cardiopulmonary bypass.

DETAILED DESCRIPTION:
Adenosine has been used for diagnosis and treatment of cardiovascular diseases for many years. New progresses in myocardial protection in the settings of acute myocardial infarction treatment put forward the its clinical use to a broader field. But the safety and effectiveness of its use in myocardial protection in the setting of open heart surgery has not been investigated intensively. Our primary results suggested that adenosine preconditioning could decrease the release of myocardial serum markers, such as cTnI. This study will focus on the safety and effectiveness of adenosine in the field of pediatric myocardial protection during surgery repair of congenital heart defects with CPB and cardioplegia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of congenital heart defects eligible for surgery treatment under cardiopulmonary bypass and cardioplegia
* Body weight less than or equals to 10kg

Exclusion Criteria:

* Cardiac surgery is performed without cardiopulmonary or cardioplegia
* Body weight more than 10Kg

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 238 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Outcome Measure: all cause mortality | within the first 30 days (plus or minus 3 days) after surgery

SECONDARY OUTCOMES:
The time of ICU stay | within the first 30 days (plus or minus 3 days) after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zhenxiao Jin, MD, Principal Investigator — Xijing Hospital
Locations (1):
- Institute of Cardiovascular Surgery, Xijing Hospital, Xi'an, Shannxi, China